CLINICAL TRIAL: NCT02469727
Title: mHealth Intervention to Promote Cancer Survivors' Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Jason Mendoza, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15563
Record Dates: First submitted 2015-06-08; First posted 2015-06-11 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Physical Activity; Quality of Life
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fitbit + Facebook (Experimental): Participants will use the Fitbit device and join the Facebook group.
  Interventions: Behavioral: Fitbit; Behavioral: Facebook group
- Usual care control (No Intervention): No intervention provided.

INTERVENTIONS:
Behavioral: Fitbit — Participants will use the FitBit device to track their physical activity
  Arms: Fitbit + Facebook
Behavioral: Facebook group — Participants will receive and post messages and receive badges on the Facebook group
  Arms: Fitbit + Facebook

SUMMARY:
The Primary Goal is to conduct a 5-10 week randomized controlled trial (RCT) of the Fitbit Flex, a popular, affordable, wearable physical activity tracking device, and the Fitbit mHealth app. The target population will be childhood cancer survivors 14-18 years old recruited from Seattle Children's Hospital. For the intervention group, peer influences will be engaged via a private, social network (e.g. a Facebook group) customized for survivors. Measurements will be completed (1) at baseline, prior to randomization, and (2) during the final week of the intervention period (follow-up measure). This study will provide initial proof of concept and allow for further customization of the intervention for childhood cancer survivors in anticipation of a future, larger proposal to study physical activity and related outcomes over a multi-year period.

ELIGIBILITY:
Inclusion Criteria:

* in remission for childhood cancer and previously treated for childhood cancer at Seattle Children's Hospital
* ≥1-year post-cancer therapy
* ambulatory without any known medical contraindications to participation
* able to complete surveys in English
* agree to install and share data from the FitBit smart phone app with the investigators

Exclusion Criteria:

* currently or previously used a wearable physical activity sensing device to improve physical activity

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Post-intervention physical activity (measured by accelerometers) | up to week 10

SECONDARY OUTCOMES:
Post-intervention health related quality of life (measured by questionnaire) | up to week 10

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States